CLINICAL TRIAL: NCT01551147
Title: A Double-blind, Placebo-controlled, Three-way Crossover Study to Compare the Safety and Efficacy of 8 Days of Therapy With ONO-6950 Versus Placebo and Montelukast (Singulair®) on Asthmatic Responses and Airway Hypersensitivity Following Allergen Challenge in Patients With Asthma
Brief Title: A Placebo and Active Controlled Study of ONO-6950 Following Allergen Challenge in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-6950POU005
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: asthma; ONO-6950; asthma in adult patients
MeSH Terms: conditions — Asthma | interventions — gemilukast; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental 200 mg dose (Experimental)
  Interventions: Drug: ONO-6950
- Active Comparator (Active Comparator)
  Interventions: Drug: Montelukast
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-6950 — 200 mg QD for 8 days
  Arms: Experimental 200 mg dose
Drug: Placebo — Placebo to match ONO-6950 tablets or over-encapsulated Montelukast tablets dosed in a similar manner
  Arms: Placebo Comparator
Drug: Montelukast — 10 mg Montelukast QD for 8 days
  Arms: Active Comparator

SUMMARY:
The primary objectives are

* to determine the effect of ONO-6950 200 mg QD versus placebo administered for 8 days on early asthmatic response (EAR) and late asthmatic response (LAR) induced by inhaled allergen
* to determine the safety and tolerability of ONO-6950 200 mg QD administered for 8 days in patients with asthma

The secondary objectives are:

* to compare the effect of ONO-6950 versus montelukast on the % decrease of FEV1 following allergen exposure, and
* to determine the effect of ONO-6950 versus placebo and montelukast on allergen-induced airway hyperresponsiveness (AHR) as measured by methacholine challenge

DETAILED DESCRIPTION:
The study will examine if ONO-6950 could alleviate EAR and LAR caused by an allergen challenge in subjects with asthma. Patients will be required to have EAR and LAR after standardized allergen challenges during the screening. Eligible patients will complete a randomized, double-blind, three-way crossover study. During each of three evaluation periods, patients will be administered either 200 mg ONO-6950, 10 mg Montelukast, or placebo for 8 days. Each evaluation period will occur over 8 days and will include various assessments following allergen challenge and methacholine challenge. The study does not require an overnight stay at the clinical research center.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, between 18 to 60 years of age, with bronchial asthma symptoms for at least 6 months
* Patients with FEV1 ≥ 70% of predicted after withholding short-acting β agonists for at least 8 hours prior to testing
* Screening allergen challenge demonstrates that the patient experiences both an early and late asthmatic response
* Sensitivity to methacholine resulting in a ≥ 20% fall in FEV1 (PC20 methacholine)
* Non-smokers with free from the usage of nicotine-containing products at least for a year prior to screening

Exclusion Criteria:

* Previous history of life-threatening asthma, respiratory tract infection and/or exacerbation of asthma within 6 weeks prior to the first screening visit
* Past or present disorders and diseases including, but are not limited to, cardiovascular, malignancy, hepatic, renal, hematological, neurological, psychiatric, endocrine, or pulmonary other than asthma
* Significant safety laboratory, ECG, or vital sign abnormalities that would place the patient at undue disk during the study procedures
* History of clinically significant multiple drug or food allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Late Asthmatic Response (3-7 hours after allergen challenge) as measured by the AUC in FEV1 | Day 7
Early Asthmatic Response as measured by the AUC in FEV1 | Day 7
Late Asthmatic Response as measured by the Maximum Fall in FEV1 | Day 7
Early Asthmatic Response as measured by the Maximum Fall in FEV1 | Day 7

SECONDARY OUTCOMES:
Differences in PC20 pre-post treatment as measured by methacholine challenge | Day 6
Differences in PC20 pre-post allergen challenge as measured by methacholine challenge | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (5):
- Canada (5):
  - Vancouver Clinical Site 530, Vancouver, British Columbia
  - Calgary Clinical Site 540, Alberta
  - Hamilton Clinical Site 550, Ontario
  - Quebec Clinical Site 510, Québec
  - Saskatoon Clinical Site 520, Saskatoon

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, FitzGerald JM, Cockcroft DW, Davis BE, Leigh R, Tanaka M, Fourre JA, Tanaka M, Nabata T, O'Byrne PM. A dual CysLT1/2 antagonist attenuates allergen-induced airway responses in subjects with mild allergic asthma. Allergy. 2016 Dec;71(12):1721-1727. doi: 10.1111/all.12987. Epub 2016 Aug 9. PMID 27444660